CLINICAL TRIAL: NCT06226064
Title: A Randomised, Double-blind, Placebo-controlled Single and Multiple Ascending Dose Study in Healthy Volunteers and Asymptomatic GRN Mutation Carriers to Investigate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VES001
Brief Title: A Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of VES001 in Healthy Participants
Acronym: SORT-IN-1
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Vesper Biotechnologies ApS (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: Ph1/VES001
Record Dates: First submitted 2023-12-07; First posted 2024-01-26 (Actual); Last update posted 2024-08-22 (Actual); Status verified 2024-08

CONDITIONS: Dementia, Frontotemporal
MeSH Terms: conditions — Frontotemporal Dementia

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- VES001 (Healthy Participants) (Experimental): Part A: Ascending single doses and Part B: Multiple ascending dose (seven days of treatment), for healthy volunteers.
  Interventions: Drug: VES001
- Placebo (Healthy Participants) (Placebo Comparator): Part A: Ascending single doses and Part B: Multiple ascending dose (seven days of treatment), for healthy volunteers.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: VES001 — VES001 is an oral, blood brain barrier penetrating ligand of sortilin.
  Arms: VES001 (Healthy Participants)
Drug: Placebo — A matching dosage form, indistinguishable from the active treatment will be used as the placebo treatment.
  Arms: Placebo (Healthy Participants)

SUMMARY:
This is a Phase 1, randomized, placebo-controlled, double-blind study to evaluate the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of single and multiple doses of VES001 in a two part followed by a multicenter, open-label Phase 1b study in asymptomatic GRN mutation carriers.

Part A will evaluate the safety, tolerability, PK, and PD of single doses of VES001 in healthy volunteers.

Part B will evaluate the safety, tolerability, PK, and PD of multiple doses of VES001 in healthy volunteers.

DETAILED DESCRIPTION:
Part A will include six cohorts, with eight participants per cohort. Participants in each cohort will be randomised in a 6:2 ratio (VES001 vs. placebo).

Part B will include three cohorts, with ten participants per cohort. Participants in each cohort will be randomised in a 8:2 ratio (VES001 vs. placebo).

ELIGIBILITY:
Inclusion Criteria Part A & B:

1. Healthy men or women aged 18 to 55 years.
2. Body Mass Index between 18 and 32 kg/m2, with a minimum weight of 50 kg.
3. Effective contraception required during the study and for at least 90 days after their last dose.
4. Participants in group 3, where the food effect is being investigated, must be able to eat a high-fat meal within 30 minutes for breakfast.

Exclusion Criteria Part A & B:

1. Medical conditions or treatments that could interfere with the study.
2. History of any known neurologic disease, cognitive impairment, or a history of seizure, (significant) head trauma, or loss of consciousness.
3. History of active malignancy (active cancer cells or tumors) within the last 5 years.
4. Abnormal laboratory test results or infectious diseases (Hepatitis B, Hepatitis C, and/or HIV).
5. Recent medication or supplement use, unless allowed by the investigator.
6. Participation in other research studies involving study treatment or devices.
7. Positive tests for illegal drugs or alcohol at screening.
8. Heavy smoking or inability to abstain from smoking during the study.
9. Excessive consumption of caffeine (more than 8 cups per day).
10. History of severe allergic reactions to medication
11. Recent blood donation or significant blood loss.
12. Pregnancy, breastfeeding, or plans to become pregnant (for women).

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 78 (Actual)
Dates: Start 2023-10-11 (Actual); Primary Completion 2024-07-26 (Actual); Study Completion 2024-07-26 (Actual)

PRIMARY OUTCOMES:
Incidence, severity, and seriousness of treatment-emergent adverse events (TEAEs). | Part A: 21 weeks. Part B: 13 weeks.
Incidence of clinically significant abnormalities in safety laboratory values. | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Pulse Rate (bpm). | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Systolic blood pressure (mmHg) and Diastolic blood pressure (mmHg). | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Electrocardiogram parameter Heart Rate (HR). | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Electrocardiogram parameter beats per minute (bpm) | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Electrocardiogram parameter PR Interval | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Electrocardiogram parameter QRS Interval | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Electrocardiogram parameter QT Interval. | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Electrocardiogram parameter QTcB (calculated using Bazzet method). | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in vital sign measurement: Electrocardiogram parameter QTcF, (calculated using Fredericia's method). | Part A: 21 weeks. Part B: 13 weeks.
Incidence of clinically significant abnormalities in physical/neurological examination findings. | Part A: 21 weeks. Part B: 13 weeks.
Change from baseline in Columbia-Suicide Severity Rating Scale (C-SSRS; Parts B). | Part A: 21 weeks. Part B: 13 weeks.

SECONDARY OUTCOMES:
Plasma PK parameter: Area under the concentration-time curve from time zero to infinity (AUCinf). | Part A: 21 weeks. Part B: 13 weeks.
Plasma PK parameter: Area under the concentration-time curve from time zero to infinity AUCinf(%extrapolated). | Part A: 21 weeks. Part B: 13 weeks.
Plasma PK parameter: Area under the concentration-time from time zero to time of last measurable concentration (AUClast). | Part A: 21 weeks. Part B: 13 weeks.
Plasma PK parameter: Apparent total clearance following extravascular administration (CL/F). | Part A: 21 weeks. Part B: 13 weeks.
Plasma PK parameter: Maximum concentration (Cmax). | Part A: 21 weeks. Part B: 13 weeks.
Plasma PK parameter: Absorption lag time (tlag). | Part A: 21 weeks. Part B: 13 weeks.
Plasma PK parameter: Time to reach maximum concentration (tmax). | Part A: 21 weeks. Part B: 13 weeks.
Plasma PK parameter: Terminal elimination half-life (t1/2). | Part A: 21 weeks. Part B: 13 weeks.
Plasma PK parameter: Apparent volume of distribution during the terminal elimination phase after extravascular administration (Vz/F). | Part A: 21 weeks. Part B: 13 weeks.
Concentration of VES001 in CSF in the highest two dose level cohorts in Part A. | Part A: 21 weeks. Part B: 13 weeks.
Concentration of VES001 in CSF in all dose level cohorts in Part B. | Part A: 21 weeks. Part B: 13 weeks.
Concentration of VES001 in plasma/CSF ratio in the highest two dose level cohorts in Part A. | Part A: 21 weeks. Part B: 13 weeks.
Concentration of VES001 in plasma/CSF ratio in all dose level cohorts in Part B. | Part A: 21 weeks. Part B: 13 weeks.
Comparison of the plasma PK of VES001 following a single oral dose in the fed and fasted state in Part A. | Part A: 21 weeks. Part B: 13 weeks.
  Refer to the PK parameters listed above.

CONTACTS AND LOCATIONS:
Overall Officials: Mads Kjolby, MD, PhD, Principal Investigator — Vesper Bio
Locations (1):
- Center for Human Drug Research, Leiden, Netherlands

IPD SHARING:
Plan to Share IPD: Undecided